CLINICAL TRIAL: NCT00445237
Title: Evaluation of the H1 Coil and H2 Coil TMS Device - Safety and Feasibility in Major Depression Episode
Brief Title: Evaluation of Deep Transcranial Magnetic Stimulation (TMS) H-Coil in the Treatment of Major Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Brainsway (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH-505
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2007-03

CONDITIONS: Major Depression
Keywords: major depression; TMS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: H1 and H2 deep TMS coils

SUMMARY:
This study is evaluating the safety and feasibility of the novel deep TMS H-coil designs in the treatment of resistant major depression in an open study using two different H-coil designs.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as suffering from treatment resistant major depression

Exclusion Criteria:

* Other axis I diagnosis
* Risk factors for convulsions
* Electroconvulsive therapy (ECT) in the last 9 months
* History of drug abuse in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-05; Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilik Levkovits, Principal Investigator — Day care hospital director
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel